CLINICAL TRIAL: NCT00033956
Title: Phase I/II Open Label Dose Escalation and Double-Blind, Placebo-Controlled Evaluation of M40403, for the Prevention of the Dose Limiting Toxicities of High Dose IV Bolus IL-2 Treatment of Metastatic Melanoma or Renal Cell Carcinoma.
Brief Title: Evaluation of M40403 for the Prevention of Dose Limiting Toxicities of High Dose IL-2
Status: Suspended | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: MetaPhore Pharmaceuticals (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: U10-01-12-002
Record Dates: First submitted 2002-04-17; First posted 2002-04-18 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2002-05

CONDITIONS: IL-2 Induced Hypotension
Keywords: Metastatic Melanoma; Renal Cell Carcinoma; IL-2; Interleukin-2; Hypotension
MeSH Terms: conditions — Melanoma; Carcinoma, Renal Cell; Hypotension | interventions — imisopasem manganese

INTERVENTIONS:
Drug: M40403

SUMMARY:
The clinical use of IL-2 is currently limited by development of dose-dependent hypotension (systolic blood pressure (SBP) < 90 mm Hg). The overall outcome is constant across sites with 20-50% of the patients requiring ICU management because of unresponsive hypotension and hyporeactivity (loss of response to vasoconstrictors). Because of the dose-limiting side effects, the duration of IL-2 dosing is frequently curtailed. Thus, hemodynamic toxicities have limited the usefulness of IL-2 therapy. M40403 has prevented both the hypotension and hyporeactivity associated with IL-2 treatment in preclinical studies. This trial will study the safety and efficacy of M40403 in the prevention or reduction of hypotension in patients receiving IL-2 therapy.

DETAILED DESCRIPTION:
High-dose interleukin-2 (IL-2) therapy is currently indicated for treatment of metastatic renal cell carcinoma and metastatic malignant melanoma, and has been associated with a 5-15% long-term clinical response. In addition, IL-2 therapy is showing promise in treatment of acute myelogenous leukemia, non-Hodgkin's lymphoma, and breast cancer, and in improving immunologic function in patients with AIDS. However, the major dose-limiting toxicity of IL-2, hypotension, severely limits the usefulness of IL-2 therapy.

Because of the unresponsive hypotension and loss of response to exogenously administered vasopressors, 20-50% of the patients receiving high dose IL-2 therapy require ICU management. These dose-limiting side effects frequently necessitate curtailing the full period of IL-2 dosing in order to reverse the hypotension and prevent subsequent renal dysfunction. Thus, hemodynamic toxicities have limited the usefulness of IL-2 therapy. A course of IL-2 therapy requires long hospitalization and intense patient monitoring during administration. As a consequence, despite favorable long-term response, few sites offer this treatment.

The availability of an agent that prevents IL-2-induced hypotension without adversely affecting the therapeutic mechanism of IL-2, would markedly facilitate IL-2 administration and at a minimum, would maximize the number of patients who could receive the full regimen of IL-2. The reduction in IL-2 toxicity may also enable higher doses and/or more frequent dosing of IL-2 to be used, with the potential of higher success of tumor response. Because M40403 may decrease the toxicity of IL-2, co-administration of M40403 may make it possible to broaden the clinical use of IL-2 to conditions where it is not currently indicated.

The indication to be studied is for use in the prevention or reduction of hypotension associated with interleukin-2 (IL-2) therapy in patients with metastatic melanoma and renal cell carcinoma.

The study is divided into a sequential dose escalation phase followed by the expansion of the selected dose in a double-blind, placebo-controlled, evaluation phase. Patients with metastatic or inoperable melanoma and renal cell carcinoma will be receiving high dose IL-2 per approved labeling as two 5-day sequences. M40403 will be administered by intravenous infusion over 30 minutes prior to each intravenous administration of high dose IL-2. Sequential panels of patients will receive increasing doses of M40403 along with IL-2 until an active dose is determined and an MTD is reached. Patients will be followed to determine the effects of M40403 on development of markers of IL-2 dose-limiting toxicity including hypotension, tachycardia, index of renal perfusion, cumulative dose of pressor required and cumulative dose of IL-2 administered. Approximately 48 patients will be studied.

ELIGIBILITY:
Inclusion Criteria:

* Patient has given signed informed consent.
* Patient has documented histologically confirmed malignant melanoma or renal cell carcinoma which is metastatic.
* Patient is eligible for high dose IV IL-2 therapy.
* Tumor dimension of at least one lesion is measurable in two dimensions.
* Patient is at least 18 years of age.
* Patient is ambulatory with good performance status (ECOG PS 0,1; Karnofsky 100-70%).
* If the patient is a woman of child bearing potential, patient is not lactating and ahs a negative pregnancy test (beta-HCG test obtained within 72 hours of enrollment) and agrees to use an adequate method of contraception for the duration of the study.
* Patient has adequate organ function as defined by:

  * WBC count >3,500 per cubic millimeter; platelet count> 100,000 per cubic millimeter;
  * Bilirubin within institutional normal range; creatinine less than or equal to 2.0 mg/dl or creatinine clearance > 50 ml/min;
  * No evidence of congestive heart failure, symptoms of coronary artery disease, serious cardiac arrhythmias or evidence of prior myocardial infarction. A pretreatment cardiac stress test must be performed within 42 days of IL-2 treatment. Patients with documented ischemia on the pretreatment cardiac stress test will be excluded from the study;
  * Adequate pulmonary reserve. Pulmonary function tests (PFTs) must be performed within 42 days of IL-2 treatment and an FEV1 > 2.0 liters or 75% of predicted for height and age is the minimum acceptable criteria for patient entry. PAtients unable to perform PFTs will be excluded from the study.
* Patient has recovered from all toxic effects of prior therapy.
* Patient has a life expectancy, in the opinion of the investigator, of at least 4 months.

Exclusion Criteria:

* Patient has an organ allograft.
* Patient has brain metastases. A Brain CT or MRI scan should be performed within 42 days of IL-2 treatment.
* Patient is know to be HIV antibody positive. HIV testing is not required for enrollment into this study.
* Patient has evidence of active infection which requires antibiotic therapy.
* Patient has received systemic corticosteroids in the four weeks prior to the first dose of study drug, or requires or is anticipated to require corticosteroids for intercurrent disease.
* Patient has received radiotherapy, chemotherapy, or immunotherapy in the four weeks prior to the first dose of study drug, or is scheduled to receive concurrent radiotherapy, chemotherapy, or immunotherapy.
* Patient has contraindication to treatment with pressor agents.
* Patient currently receives chronic medication for asthma.
* Patient has a history of another malignancy other than basal cell skin cancer within 5 years prior to the first dose of study drug.
* Patient has any significant medical disease other than the malignancy which, in the opinion of the investigator, may interfere with completion of the study.
* Patient has previously received any IL-2 therapy.
* Patient has received another investigational medication within 4 weeks prior to M40403 administration or is scheduled to receive an investigational drug other than M40403 during the course of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48
Dates: Start 2001-12

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Northwestern University Medical School, Chicago, Illinois
  - Providence Portland Medical Center, Portland, Oregon
  - Huntsman Cancer Institute, Salt Lake City, Utah